CLINICAL TRIAL: NCT01358786
Title: Seroma at the Donor Site of the TRAM Flap, With or Without Quilting Suture.
Brief Title: Seroma at the Donor Site of the TRAM Flap, With or Without Quilting Suture: A Comparative Study Using Ultrasound
Acronym: STRAMQUSG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Graduate Program in Plastic Surgery, School of Medicine, Luis Antonio Rossetto
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CEP 1995 08; CEP 1995/08 (Other: Comisão de Ética Médica do Hospital São Paulo)
Record Dates: First submitted 2011-05-16; First posted 2011-05-24 (Estimated); Last update posted 2011-05-26 (Estimated); Status verified 2009-06

CONDITIONS: Seroma
Keywords: Quilting suture; seroma; Procedure; Surgery
MeSH Terms: conditions — Seroma

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- no quilting sutures but drains (No Intervention)
  Interventions: Procedure: quilting suture
- quilting sutures and drains (Experimental)
  Interventions: Procedure: quilting suture
- quilting sutures but no drains (Experimental)
  Interventions: Procedure: quilting suture

INTERVENTIONS:
Procedure: quilting suture — * quilting sutures and drains
  * quilting sutures but no drains
  Other Names: points

SUMMARY:
Patient undergoing breast reconstruction with lower abdominal flap, benefit when points are used for membership (between the aponeurosis of the abdominal flap and underlying muscles) for closing the donor area, where there is reduced incidence of complications.

DETAILED DESCRIPTION:
This study evaluated seroma formation at the donor site of the TRAM patients who underwent breast reconstruction. Forty-eight breast reconstructions were performed using the bipedicled TRAM flap. The patients were randomly allocated into three groups of 16 participants each: DN group, use of suction drains but no quilting sutures between the remaining abdominal flap and musculoaponeurotic layer of the anterior abdominal wall; QS+DN group, use of quilting sutures and suction drains; and QS group, use of quilting sutures but no suction drains. In order to determine seroma formation, ultrasound examinations were performed on postoperative days 7 and 14 in 5 regions of the abdominal wall: epigastric, umbilical, hypogastric, right iliac, and left iliac regions.

ELIGIBILITY:
Inclusion Criteria:

* were age between 20 and 65 years
* body mass index (BMI) ≤ 30 kg/m2
* non-smokers.

Exclusion criteria:

* no skin excess in the infraumbilical region
* previous abdominoplasty
* uncontrolled systemic disease
* such as diabetes mellitus and arterial hypertension
* collagen diseases
* psychiatric disorders
* large weight loss
* and/or postoperative abdominal scars that could hinder flap vascularization.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Reducing seroma in donor site of the TRAM flap | 15 days
  Seroma formation was identified clinically and confirmed by ultrasound examination. Clinical examination consisted of evaluation of early symptoms (bulging and distension of the skin, signs of fluid accumulation), palpation, and percussion. Ultrasound examination was performed on postoperative days 7 and 14 to detect the presence of seroma at the TRAM flap donor site. The patients were placed in the supine position during the examination. Upon detection of seroma, ultrasound-guided puncture was performed, and the number of punctures and volume of seroma aspirated were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: luis Rossetto, MD, Study Director — Graduate Program in Plastic Surgery, School of Medicine, Universidade Federal de São PaConception and design of the study, drafting the article, revising it critically for important intellectual content, and final approval of the version to be submitted.

REFERENCES:
- [Background] 1. Hartrampf CR, Jr, Scheflan M, Black PW. Breast reconstruction with a transverse abdominal island flap. Plast Reconstr Surg. 1982;69:216-225. 2. Andrades P, Prado A, Danilla S, et al. Progressive tension sutures in the prevention of postabdominoplasty seroma: a prospective, randomized, double-blind clinical trial. Plast Reconstr Surg. 2007;120:935-946. 3. Baroudi R, Ferreira CA. Contouring the hip and the abdomen. Clin Plast Surg. 1996;23:551-572. 4. Rossetto LA, Garcia EB, Abla LF, Neto MS, Ferreira LM. Quilting suture in the donor site of the transverse rectus abdominis musculocutaneous flap in breast reconstruction. Ann Plast Surg. 2009;62:240-243. %. Di Martino M, Nahas FX, Barbosa MV, et al. Seroma in lipoabdominoplasty and abdominoplasty: a comparative study using ultrasound. Plast Reconstr Surg. 2010;126:1742-1751.
- [Derived] Rossetto LA, Garcia EB, Abla LE, Ferreira LM. Seroma and quilting suture at the donor site of the TRAM flap in breast reconstruction: a prospective randomized double-blind clinical trial. Ann Plast Surg. 2014 Apr;72(4):391-7. doi: 10.1097/SAP.0b013e3182610b11. PMID 23407260
- See also: Federal University of Saint Paul — http://www.unifesp.br